CLINICAL TRIAL: NCT00090870
Title: A Phase II Study Of Peg-Intron, GM-CSF And Thalidomide In Metastatic Renal Cell Carcinoma
Brief Title: PEG-Interferon Alfa-2b, Sargramostim, and Thalidomide in Treating Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical collaborator pulled funding.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000378049; MUSC-100614; CELGENE-MUSC-100614; MUSC-HR-10423
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — peginterferon alfa-2b; Granulocyte-Macrophage Colony-Stimulating Factor; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-Intron, BM-CSF and thalidomide (Experimental)
  Interventions: Biological: PEG-interferon alfa-2b; Biological: GM-CSF; Drug: thalidomide

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Peg-Intron 1ug/kg Subcutaneous on day 1 and day 8 of each cycle. Each cycle is 21 days.
Biological: GM-CSF — GM-CSF 250 ug/m2 subcutaneously daily from days 1-10 or each 21 day Peg-Intron cycle
Drug: thalidomide — 200mg daily by mouth

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining PEG-interferon alfa-2b with sargramostim and thalidomide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving PEG-interferon alfa-2b together with sargramostim and thalidomide works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response to PEG-interferon alfa-2b, sargramostim (GM-CSF), and thalidomide in patients with metastatic renal cell carcinoma.

Secondary

* Determine duration of response in patients treated with this regimen.
* Determine the tolerance to and toxicity of this regimen in these patients.
* Determine the median and progression-free survival of patients treated with this regimen.

OUTLINE: Patients receive PEG-interferon alfa-2b subcutaneously (SC) on days 1 and 8, sargramostim (GM-CSF) SC on days 1-10, and oral thalidomide once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Metastatic disease
* Measurable disease

  * Unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan or MRI

    * Histologic confirmation required if measurable disease is confined to a solitary lesion
  * The following are not considered measurable disease:

    * Bone disease only
    * Pleural or peritoneal metastases
    * CNS lesions
    * Irradiated lesions unless disease progression was documented after prior radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* No decompensated liver disease

Renal

* Creatinine ≤ 2.0 mg/dL

Immunologic

* No known or suspected hypersensitivity to interferon alfa or to any excipient or vehicle included in the formulation or delivery system
* No history of autoimmune disease
* No autoimmune hepatitis
* No immunosuppressed transplantation recipients

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception 4 weeks before, during, and for 4 weeks after study participation
* No pre-existing thyroid abnormalities for which thyroid function cannot be maintained in the normal range
* No severe psychiatric condition or disorder, including suicidal ideation or attempt
* No other active malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzair B. Chaudhary, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To define the response rate in metastatic renal cell carcinoma patients receiving Peg-Intron, GM-CSF and thalidomide
Time Frame: while on study, every 4 cycles; while off study, every 3 months for 1 year, then every 6 month for 2 years, then every year
Population: Data for this endpoint was not collected
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Time Frame: time from registration to the time of progressive disease among patients who achieve at least a partial response to treatment.
Population: Data for this endpoint was not collected
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency of Adverse Events Assessed by NCI CTC Version 2
Time Frame: From the first day of treatment until the end of treatment visit, an average of 6 months
Population: Data for this endpoint was not collected
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: From registration until diease progression or death, whichever comes first.
Population: Data for this endpoint was not collected
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From day 1 of study treatment until end of study, for an average of 6 months
Description: Data for this endpoint was not collected
Arm/Group | PEG-Intron, BM-CSF and Thalidomide
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes